CLINICAL TRIAL: NCT05265260
Title: Barriers to Early Progress in Cochlear Implant Outcomes: a Non-interventional Feasibility Study
Brief Title: Factors Affecting Early Progress of Cochlear Implant Outcomes in Adults
Acronym: PROGRESS
Status: Completed | Type: Observational
Sponsor: Cochlear (Industry)
Collaborators: EVAMED (Other)
Responsible Party: Sponsor
Other Study IDs: EMEA5798
Record Dates: First submitted 2022-02-23; First posted 2022-03-03 (Actual); Results first posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2023-10

CONDITIONS: Sensorineural Hearing Loss, Bilateral
Keywords: Cochlear implant; Sentence recognition; Cognitive processing; Electrophysiology
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to understand how audiometric, cognitive and electrophysiological results relate to sentence recognition score in adults using currently a Nucleus cochlear implant.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects, 18 years or older
* Subjects unilaterally implanted or bilaterally implanted with at least 6 months separating the two cochlear implantations.
* Subjects who have been implanted between January 2016 and December 2021.
* Subjects have received a Nucleus CI: CI512, CI522 or CI532 cochlear implants with non-rotating magnet, or CI600 series equivalent CI612, CI622 and CI632 with rotating magnet and external sound processors CP900 or CP1000 behind-the-ear, or Kanso or Kanso 2 off-the-ear types.
* Subjects who are fluent in French (language used in the questionnaire and speech tests)
* Subjects who are not opposed to participating in the study
* Subjects for who the medical record data is available throughout the defined data search period.

Exclusion Criteria:

* Subjects with single-sided deafness (SSD).
* Subjects who are not affiliated to the French Social Security.
* Subjects who are under legal protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Cochlear Implants recipients who are using currently a Nucleus cochlear implant with moderately severe to profound bilateral sensorineural hearing loss.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu Marx, MD, Principal Investigator — Hôpital Pierre-Paul Riquet
Locations (1):
- Hôpital Pierre-Paul Riquet, ORL, otoneurologie et ORL pédiatrique, Toulouse, France

IPD SHARING:
Plan to Share IPD: No
Cochlear do not have an approved platform for public sharing of IPD collected in this study. Data may be provided to individual researchers on request

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 32 participants were recruited between 21 April 2022 and 24 August 2022. The aim was to recruit 30 participants with data for the primary endpoint. As it was noted during the data collection period that data was missing, the number was increased to 32.
Groups:
- Adults Using Currently a Nucleus Cochlear Implant: Adults (>18 years) unilaterally implanted or bilaterally implanted with at least 6 months separating the two cochlear implantations.
Period: Overall Study
Arm/Group | Adults Using Currently a Nucleus Cochlear Implant
Started | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Adults Using Currently a Nucleus Cochlear Implant
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.0 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex/ gender information has not been collected.
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race information has not been collected.
Region of Enrollment [Number; unit: participants]
  France | 32

OUTCOME MEASURES:

1. Primary Outcome: Score of the French MBAA2 Sentence Recognition Test in Quiet
Description: Participants are classified in good or poor performer based on the score of the French MBAA2 sentence recognition test. A good performer has a score of ≥90/100 correct sentence. A bad performer has a score of <90/100 correct sentence.
Time Frame: 1 month post activation
Measure: Count of Participants; unit: Participants
Arm/Group | Adults Using Currently a Nucleus Cochlear Implant
Number analyzed (Participants) | 32
Participants
  Good performer | 13
  Bad performer | 19

ADVERSE EVENTS:
Description: Deaths, serious adverse events and non-serious adverse events were not assessed.
Arm/Group | Adults Using Currently a Nucleus Cochlear Implant
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-20): https://cdn.clinicaltrials.gov/large-docs/60/NCT05265260/Prot_SAP_000.pdf